CLINICAL TRIAL: NCT04263974
Title: Effectiveness of a Mobile Application of Exercise and Education for the Management of Patients With Hand Osteoarthritis and Rheumatoid Arthritis on Self-reported Functional Ability, Dexterity, Pinch and Grip Strength, Pain Intensity and Stiffness
Brief Title: Effectiveness of an Exercise Program and Education Through a Mobile Application for the Management of Patients With Hand Osteoarthritis and Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Fundación Pública Andaluza Progreso y Salud (Other); Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Principal Investigator, Alberto Marcos Heredia-Rizo, Assistant Professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI_RH_2018
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Rheumatoid Arthritis - Hand Joint; Osteoarthritis Hand; Pain; Mobility Limitation; Stiffness of Hand, Not Elsewhere Classified
MeSH Terms: conditions — Pain; Mobility Limitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone Application (Experimental): A protocol of exercises and general recommendations based on the current scientific evidence will be provided through a smartphone application. A follow-up of the use of the application will be carried out. The treatment protocol will last 6 months, during which a minimum of 4 weekly sessions of exercises will be carried out at home.
  Each pathology will have an unique program of exercises and recommendations.
  Interventions: Other: Smartphone Application
- Conventional Treatment (Active Comparator): Those in this group will received the conventional treatment protocol provided within the Andalusian Public Health System. This will consist on the delivery of an exercise program and recommendations using a sheet of paper. Participants will be told to perform the exercises during 6 months, with minimum of 4 weekly sessions of exercise that will be carried out at home.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Smartphone Application — Exercises and recommendations, based on current scientific evidence, and delivered through the app for Smartphone called CareHand. The intervention protocol is based on strengthening and stretching recommendations for rheumatoid arthritis and osteoarthritis in hands, transferred to an application format through explanatory videos together with tools to improve the autonomy, motivation and adherence of the patient
  Arms: Smartphone Application
Other: Conventional treatment — Conventional approach provided by the Andalusian Public Health System in Primary Care settings. This approach consists of routine visits to the general practitioner specialist, and the delivery of an exercise sheet and recommendations. This general mobility and stretching worksheet contains detailed images, as well as a description of how to perform the exercises and the dose to be taken. While most exercises are intended for the wrist and hands, this sheet also includes basic exercises for the elbow joint.
  Arms: Conventional Treatment

SUMMARY:
Strengthening and stretching exercise programs, and recommendations to protect the affected joint have shown to be effective both clinically and economically in conditions such as hand osteoarthritis and hand rheumatoid arthritis. However, their application format is not up to date. In this sense, problems such as the lack of monitoring by the health professional and the lack of patients motivation may cause poor adherence to the treatment protocol, which is one of the main predictors of treatment efficiency. Therefore, an smartphone application has been developed for the rehabilitation of hand osteoarthritis and rheumatoid arthritis to enhance patients adherence and motivation. The smartphone application includes: a) exercise programs and recommendations based on the most up to date scientific evidence adapted to the pathology; and b) enhancers of patient adherence to treatment (patient diaries and behavioral change strategies).The objective is to develop a cost effective digital solution to optimize the health care offered to these pathologies based on up to date scientific evidence in order to improve the functional ability and the quality of life of these patients, and to reduce the number of consultations to primary and specialized care.

ELIGIBILITY:
Inclusion Criteria:

1. Hand Osteoarthritis (OA) patients:

   * Subjects with hand osteoarthritis according to the American College of Rheumatology (ACR) classification criteria for clinical OA; hand pain, aching or stiffness and 3 of the following points;

     1. Hard tissue enlargement of 2 or more of 10 hand joints.
     2. Hard tissue enlargement of 2 or more interphalangeal joints.
     3. Fewer than 3 swollen Metacarpal joints.
     4. Deformity of 1 or more of 10 hand joints.
   * Pain and dysfunction in the joints of the hands and/or wrists
   * Possession of a smartphone with internet.
2. Rheumatoid Arthritis (RA) Hand patients:

   * Subjects with hand arthritis according to the American College of Rheumatology (ACR) clinical and immunological criteria for clinical RA. Patients must meet 4 of the following seven criteria:

     1. Morning stiffness in and around joints lasting at least 1 hour.
     2. Swelling in three or more joints.
     3. Swelling in hand or wrist joints,
     4. Symmetrical joint swelling.
     5. erosions or decalcification on radiographs of hand and/or wrist.
     6. Rheumatoid nodules.
     7. Abnormal serum rheumatoid factor.
   * Pain and dysfunction in the joints of the hands and/or wrists.
   * Possession of a smartphone with internet

Exclusion Criteria:

1. Hand Osteoarthritis Patients:

   * Age under 18 years
   * People with cognitive impairment
   * Surgery on any upper limb joint or fracture in the upper limb within the previous 6 months
   * People on the waiting list for upper limb surgery.
   * Persons who have received steroid injections into the joints of their hands in the two months prior to recruitment.
   * People with inflammatory rheumatic disease (arthritis, spondylitis or cancer)
2. Rheumatoid Arthritis Hand Patients

   * Age under 18 years
   * People with cognitive impairment
   * Surgery on any upper limb joint or fracture in the upper limb within the previous 6 months
   * People on the waiting list for upper limb surgery.
   * Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Self reported functional ability assessed using Michigan Hand Questionnaire (MHQ) in patients with hand Rheumatoid Arthritis | Change from Baseline Michigan Hand Questionnaire (MHQ) at 3 and 6 months
  An outcome measurement tool specifically for chronic hand conditions providing information on functionality, satisfaction, appearance and perceived pain, with 37 questions divided into 6 subscales
Self reported functional ability assessed by Australian/Canadian (AUSCAN) Osteoarthritis Hand Index in patients with Hand Osteoarthritis | Change from Baseline Australian/Canadian (AUSCAN) Osteoarthritis Hand Index at 3 and 6 months
  A self administered measure to assess hand pain, stiffness and functionality in persons with hand osteoarthritis

SECONDARY OUTCOMES:
Grip strength assessed using a hydraulic grip dynamometer | Change from Baseline Grip Strength at 3 months
  The Maximun power of the hand muscles used to firmly grasp an object by wrapping the fingers around it, pressing it against the palm, and using the thumb to apply counter-pressure, using a Hydraulic grip dynamometer
Pinch strength assessed using a hydraulic pinch dynamometer | Change from Baseline Pinch strength at 3 months
  The maximun power of the pinch muscles, pressing the tip thumb against the tip index finger, using an Hydraulic pinch dynamometer
Self reported pain assessed using a Visual Analog Scale of pain | Change from Baseline Visual Analog Scale of Pain at 1, 3 and 6 months
  Amount of perceived pain represented on a scale of 0 (no pain) to 10 (worst pain)
Self reported stiffness assessed using a Visual Analog Scale of Stiffness | Change from Baseline Visual Analog Scale of Stiffness at 3 and 6 months
  Amount of perceived stiffness represented on a scale of 0 (no stiffness) to 10 (worst stiffness)
Self-reported functional ability assessed by QuickDASH Questionnaire | Change from Baseline QuickDASH Questionnaire at 1, 3 and 6 months
  Short form of the Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire. A self administered outcome tool designed to measure physical function and symptoms in persons with musculoskeletal disorders of the upper limb
Dexterity assessed using the Nine Hole Peg Test | Change from Baseline Nine Hole Peg Test at 3 months
  Plastic instrument woth a shallow round dish to contain pegs and nine holes on the opposite side. Consist of measuring the time spent to place and remove all the pegs from the holes.
Quality of life assessed using the EQ-5D-5L questionnaire | Change from Baseline EQ-5D-5L Questionnaire at 3 and 6 months
  A brief multi-attribute health status measure divided in five dimensions questions with Likert response options and a visual analog scale of Health
Economic factors relating to cost-utility | Change from Baseline Economic factors relating to cost-utility at 6 months
  Absence due to illness, absence from unpaid work, use of health resources (number of consultations to primary care, specialist doctor, physical therapy, occupational therapy, emergency department), pharmacological use for the pathology, medical or technical equipment purchased for the pathology

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez Sanchez-Laulhe P, Luque-Romero LG, Barrero-Garcia FJ, Biscarri-Carbonero A, Blanquero J, Suero-Pineda A, Heredia-Rizo AM. An Exercise and Educational and Self-management Program Delivered With a Smartphone App (CareHand) in Adults With Rheumatoid Arthritis of the Hands: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2022 Apr 7;10(4):e35462. doi: 10.2196/35462. PMID 35389367
- [Derived] Rodriguez-Sanchez-Laulhe P, Luque-Romero LG, Blanquero J, Suero-Pineda A, Biscarri-Carbonero A, Barrero-Garcia FJ, Heredia-Rizo AM. A mobile app using therapeutic exercise and education for self-management in patients with hand rheumatoid arthritis: a randomized controlled trial protocol. Trials. 2020 Sep 10;21(1):777. doi: 10.1186/s13063-020-04713-4. PMID 32912305